CLINICAL TRIAL: NCT06828757
Title: A Phase III Prospective, Randomized, Parallel-Controlled Clinical Study of Nanocrystalline Megestrol in Malnourished Patients With First-Line Non-Small Cell Lung Cancer
Brief Title: Clinical Study of Nanocrystalline Megestrol in Malnourished Patients With First-Line Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NM2025
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Treatment cohort
  Interventions: Drug: nanocrystalline megestrol oral suspension + PD-1/L1 inhibitor combined with chemotherapy
- Cohort 2 (Experimental): Control cohort
  Interventions: Drug: PD-1/L1 inhibitor combined with chemotherapy

INTERVENTIONS:
Drug: nanocrystalline megestrol oral suspension + PD-1/L1 inhibitor combined with chemotherapy — Oral suspension of nanocrystalline megestrol is taken orally once a day until disease progression or 12 weeks (maximum duration of 12 weeks) PD-1/L1 inhibitors combined with chemotherapy are given every 3 weeks for one dosing cycle.
  Arms: Cohort 1
Drug: PD-1/L1 inhibitor combined with chemotherapy — PD-1/L1 inhibitors combined with chemotherapy are given every 3 weeks for one dosing cycle.
  Arms: Cohort 2

SUMMARY:
This prospective interventional clinical study evaluates the efficacy of nanocrystalline megestrol combined with standard care in improving appetite and weight compared to standard care alone in first-line treatment of NSCLC.

DETAILED DESCRIPTION:
For patients with locally advanced or metastatic NSCLC who are not eligible for curative treatment-including those with non-squamous cell carcinoma harboring EGFR wild-type and ALK fusion-negative status-there remains a lack of evidence-based data on the association between improving high-risk malnutrition (NRS2002 score ≥3) and clinical benefit. Additionally, clinical research on nanocrystalline megestrol, a novel megestrol formulation, in the Chinese population is limited. Furthermore, data on its use in the first-line treatment of high-risk NSCLC with standard care are scarce. Integrating nanocrystalline megestrol into antitumor therapy to address malnutrition, enhance appetite, and promote weight gain represents a clinically meaningful and feasible approach. This strategy holds promise for improving quality of life while addressing the critical issue of survival benefit.

ELIGIBILITY:
Inclusion Criteria:

* (1) Voluntarily sign a written ICF. (2) The age at the time of enrollment is ≥18 years old. (3) The physical fitness score of Eastern Tumor Cooperation Organization (ECOG) is 0-2.

  (4) The expected survival period is ≥6 months. (5) According to the 8th edition of the TNM stage classification of lung cancer with histological or cytologic evidence that cannot undergo complete surgical resection and cannot undergo radical synchronous/sequential chemoradiation and treatment ( ⅢB/ⅢC phase), metastatic (IV phase) NSCLC.

  (6) The subject has not received systemic chemotherapy for locally advanced or metastatic NSCLC. For patients who have received adjuvant/radiotherapy, neoadjuvant/radiotherapy or radical chemotherapy for locally advanced diseases, if the disease progression occurs after the end of the last treatment> After 6 months, you are eligible to participate in this study.

  (7) Subjects who had previously received PD-1/L1 inhibitors in the neoadjuvant stage were allowed to participate in this study after the investigator's evaluation and consent. Participants who had received PD-1/L1 inhibitors in the adjuvant stage or in the consolidation treatment stage after radical chemoradiotherapy were not allowed to participate in this study.

  (8) No EGFR-sensitive mutation or ALK gene translocation changes. For scaly NSCLC subjects with a history of smoking or who are still smoking, they are considered negative if the previous EGFR and ALK status are unknown.

  (9) There is at least one measurable lesion according to RECIST v1.1, and the lesion is suitable for repeated and accurate measurement.

  (10) There is a high risk of malnutrition (nutrition risk screening 2002 score ≥3 points); (11) Determine good organ functions through the following requirements:

  a) Hematology (no blood components and cell growth factor support therapy were used within 7 days before the start of the study): i. Absolute neutrophil value ANC ≥ 1.5 × 109/L (1,500/mm3); ii.Platelet count ≥ 100 × 109/L (100,000/mm3); iii.Hymoglobin ≥ 90 g/L. b) Kidney: i. Creatinine clearance* (CrCl) Calculated value ≥ 50 mL/min

  * The Cockcroft-Gault formula will be used to calculate CrCl (Cockcroft-Gault formula) CrCl (mL/min) = {(140 Age) × Weight (kg) × F/ (SCr (mg/dL) × 72) F=1 for males; F=0.85 for females; SCr = serum creatinine. ii. Urine protein ≤1 or 24 hours (h) Urine protein quantification < 1.0 g. c) Liver: i. serum total bilirubin (TBil) ≤ 1.5 × ULN; for patients with liver metastasis or evidence-confirmed/suspected Gilbert disease, TBil ≤ 3 × ULN ii. AST and ALT ≤ 2.5 × ULN; for patients with liver metastasis or evidence-confirmed/suspected Gilbert disease, TBil ≤ 3 × ULN; for patients with AST and ALT ≤ 2.5 × ULN; for patients with liver Metastatic patients, AST and ALT ≤ 5× ULN iii. Serum albumin (ALB) ≥28 g/L d) Coagulation function: i. International standardized ratio and activated partial thromboplastin time ≤ 1.5 × ULN (unless the patient is receiving anticoagulant treatment and the coagulation parameters (PT/INR and APTT) at screening are within the expected range of treatment with anticoagulant).

  e) Cardiac function: i. Left ventricular ejaculation fraction (LVEF) ≥50%. (12) Female patients with fertility must undergo urine or serum pregnancy test within 3 days before the first medication (if the urine pregnancy test result cannot be confirmed to be negative, serum pregnancy test is required, and the serum pregnancy result shall prevail), and The result was negative. If a female patient with fertility has sex with an unsterilized male partner, the patient must adopt an acceptable contraceptive method from screening and must agree to the contraceptive method for continuous use within 120 days of the last dose of the study drug; Whether to stop contraceptive after this time point should be discussed with the researchers. If a male patient who is not sterilized has sex with a female partner with fertility, the patient must adopt an effective contraceptive method from the beginning of screening to the 120th day after the last dose; as to whether contraceptive is stopped after this time point, the patient should use the following: Researcher discussion.

  (13) The patient is willing and able to comply with the visits, treatment plans, laboratory tests specified in the schedule, and comply with other research requirements.

Exclusion Criteria:

* (1) NSCLC diagnosed with EGFR sensitivity mutation or ALK gene translocation; Histologic presence of a small cell carcinoma component is not allowed to enroll.

  (2) Presence of dysphagia, malabsorption or uncontrollable vomiting and any other condition that affects gastrointestinal absorption; Ongoing tube feeding or parenteral nutrition; Presence of anorexia nervosa, anorexia due to psychiatric disorders, or pain that makes it difficult to eat.

  (3) Is taking or plans to take other appetite or weight increasing drugs, such as: adrenal corticosteroids (except for short-term use of dexamethasone during chemotherapy), androgens, progesterones, thalidomide, olanzapine, and anamolin or other appetite stimulants.

  (4) Patients with Cushing's syndrome, adrenal or pituitary insufficiency; Difficult to control diabetes patients.

  (5) Current imaging or clinical manifestations of gastrointestinal obstruction. (6) Active autoimmune disease requiring systemic therapy within the past two years (such as treatment with disease-modifying drugs, corticosteroids, immunosuppressants). Previous history of non-infectious pneumonitis/interstitial lung disease requiring systemic glucocorticoid therapy or current presence of non-infectious pneumonitis.

  (7) Current presence of uncontrolled comorbid diseases, including but not limited to decompensated cirrhosis, renal failure, uncontrolled metabolic disorders, severely active peptic ulcer disease, or gastritis, or psychiatric illness/social conditions that would limit the patient's compliance with study requirements or affect the patient's ability to provide written informed consent.

  (8) Unstable angina, myocardial infarction, congestive heart failure (grade 2 and above determined by the functional classification of the New York Heart Association) or vascular disease (such as aortic aneurysm with risk of rupture) requiring hospitalization within 12 months prior to the first dose, or other cardiac damage that may affect the safety evaluation of the study drug (such as poorly controlled arrhythmia, myocardial ischemia); History of esophageal and gastric varices, severe ulcers, gastrointestinal perforation and/or fistulas, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), intra-abdominal abscess, or acute gastrointestinal bleeding within 6 months prior to the first dose.

  (9) Any arterial thromboembolic event within 6 months prior to the first dose, venous thromboembolic event of NCI CTCAE version 5.0 grade 3 and above (requiring urgent medical intervention, such as pulmonary embolism or intracavenital embolism), transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy; Acute exacerbation of chronic obstructive pulmonary disease within 1 month prior to the first dose; Current hypertension with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg after treatment with oral antihypertensive medications.

  (10) Have a history of severe bleeding tendency or coagulation dysfunction; Significant clinically significant bleeding symptoms within 1 month prior to the first dose, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or coughing up ≥1 teaspoon of fresh blood or small blood clots or only coughing up blood without sputum, patients with blood in sputum are allowed to be enrolled), nasal bleeding (excluding epistaxis bleeding and retracting rhinoblood).

  (11) Serious infection within 4 weeks prior to the first dose, including but not limited to comorbidities requiring hospitalization, sepsis or severe pneumonia; Active infection (excluding antiviral therapy for hepatitis B or C) that has received systemic anti-infective therapy within 2 weeks prior to the first dose.

  (12) Any previous or current disease, treatment, or laboratory abnormality that may confound the results of the study, affect the patient's full participation in the study, or may not be in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Appetite improvement level | Time from first subject dose to study completion, or up to 36 month
  Proportion of subjects with an improvement in appetite based on A/CS-12 during the treatment period; (An increase of ≥4 points or ≥37 points on the A/CS-12 scale is defined as an improvement in appetite)
Weight improvement level | Time from first subject dose to study completion, or up to 36 month
  Proportion of subjects with an increase from baseline in BMI during the treatment period.

SECONDARY OUTCOMES:
progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  defined as the duration from the start treatment to progression, or patient death
Objective Response Rate (ORR) | Time from first subject dose to study completion, or up to 36 month
  define as the proportion of subjects who have a complete response (CR) or a partial response (PR)
L3 SMI | Time from first subject dose to study completion, or up to 36 month
  Changes in L3 skeletal muscle index (L3 SMI).
Nutritional status improvement level | Time from first subject dose to study completion, or up to 36 month
  Assess the patient's nutritional improvement from treatment based on the Nutritional Risk Screening Score Short Form (NRS2002)
The number of cycles of treatment completed | Time from first subject dose to study completion, or up to 36 month
  Number of cycles from the start of the first treatment to the completion of the treatment
The occurrence of treatment reduction | Time from first subject dose to study completion, or up to 36 month
  Proportion of the number of patients with treatment reduction to the total number of patients from the first treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China